CLINICAL TRIAL: NCT02969005
Title: Use of a Radiopaque Localizer Grid and Methylene Blue Staining as an Aid to Reduce Radiation Exposure in Resection Small Femur Lesions
Brief Title: Use of a Radiopaque Localizer Grid and Methylene Blue Staining as an Aid to Reduce Radiation Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Guoxin Nan, Director, Children's Hospital of Chongqing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChongqingMUCH
Record Dates: First submitted 2016-10-24; First posted 2016-11-21 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Bone Diseases
Keywords: radiopaque localizer grid; methylene blue; reduce radiation exposure
MeSH Terms: conditions — Bone Diseases | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgery group (Experimental): The dissection was continued into the deeper layers until the bone lesion was visualized, and the bone lesion was then thoroughly resected.
  Interventions: Radiation: surgical treatment

INTERVENTIONS:
Radiation: surgical treatment — Use of a radiopaque localizer grid and methylene blue staining as an aid to resect the lesions

SUMMARY:
Localization of small femur lesions for resection can be challenging and may be associated with the need for significant fluoroscopic imaging and tissue dissection.

DETAILED DESCRIPTION:
This study was performed to evaluate the use of a radiopaque localizer grid along with methylene blue staining for resection of small femur lesions in children, and to determine this technique's effectiveness at reducing radiation exposure and tissue injury.

ELIGIBILITY:
Inclusion Criteria:

* patients with lesions <20.0 mm

Exclusion Criteria:

* patients with lesions >20.0 mm

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The times of C-arm fluoroscopy used | intraoperative

SECONDARY OUTCOMES:
incision length | intraoperative

IPD SHARING:
Plan to Share IPD: No